CLINICAL TRIAL: NCT04068532
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, 2-Period, 2-Sequence Crossover Study to Explore Pharmacodynamic Effects of BIIB104 on Brain Circuitry Using BOLD Functional MRI and Arterial Spin Labeling in Healthy Participants
Brief Title: A Study to Explore Pharmacodynamic Effects of BIIB104 on Brain Circuitry in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 263HV101; 2019-001104-38 (EudraCT Number)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive matching placebo to BIIB104 on Days 1-4 in treatment periods 1 or 2.
  Interventions: Drug: Placebo
- BIIB104 (Experimental): Participants will receive BIIB104 on Days 1-4 in treatment periods 1 or 2.
  Interventions: Drug: BIIB104

INTERVENTIONS:
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo
Drug: BIIB104 — Administered as specified in the treatment arm.
  Arms: BIIB104

SUMMARY:
The primary objective of the study is to explore the pharmacodynamic (PD) effects of BIIB104 on brain circuitry associated with emotional processing in healthy participants.

The secondary objectives of the study are to evaluate the safety and tolerability of BIIB104 in healthy participants; To further explore the PD effects of BIIB104 on brain circuitry associated with emotional processing in healthy participants; To explore the PD effects of BIIB104 on brain circuitry associated with working memory in healthy participants using the N-Back; To explore the PD effects of BIIB104 on regional cerebral blood flow (CBF) in healthy participants; To explore the PD effects of BIIB104 on brain circuitry during resting state in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2), inclusive.
* Right-handed as determined by the Edinburgh Handedness Inventory (score of >40) [Oldfield 1971].

Key Exclusion Criteria:

* Previous participation in this study or previous studies with BIIB104.
* Body weight <55 kg.
* History of severe allergic or anaphylactic reactions, or systemic hypersensitivity reaction to BIIB104 or any allergic reactions that in the opinion of the Investigator are likely to be exacerbated by any component of the study treatment.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Faces Versus Shapes Emotional Faces Task Blood Oxygen Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Contrasts to Day 4 Within a Priori Defined Regions of Interest | Baseline, Day 4

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening up to Day 44
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death, in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event), however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.
Change From Baseline in Emotional Faces Task Blood Oxygen Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Contrasts to Day 1 and Day 4 Within a Priori Defined Regions of Interest | Baseline, Day 1, Day 4
Change From Baseline in N-Back Task Blood Oxygen Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Contrasts to Day 1 and Day 4 Within a Priori Defined Regions of Interest | Baseline, Day 1, Day 4
Change From Baseline in Arterial Spin Labeling (ASL)-Derived Maps of Regional Cerebral Blood Flow (CBF) at Rest to Day 1 and Day 4 Within a Priori Defined Regions of Interest | Baseline, Day 1, Day 4
Change From Baseline in Blood Oxygen Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI)-Derived Intrinsic Functional Connectivity Networks at Rest to Day 1 and Day 4 Within a Priori Defined Regions of Interest | Baseline, Day 1, Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/